CLINICAL TRIAL: NCT07240389
Title: Evaluation of Therapeutic Outcomes in Vulvar Lichen Sclerosus Treated With Corticosteroids, Calcineurin Inhibitors, and Platelet-rich Plasma (PRP).
Brief Title: Treatment of Vulvar Lichen Sclerosus With Corticosteroid Ointment, Calcineurin Inhibitor Ointment, and Platelet-Rich Plasma (PRP) Therapy.
Acronym: VULIS-3T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milosz Pietrus (Other)
Responsible Party: Sponsor-Investigator, Milosz Pietrus, MD PhD, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UJ/2025/VULIS-3T; N41/DBS/001550 (Other Grant/Funding Number: Jagiellonian University Collegium Medicum)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: Vulvar Lichen Sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Therapeutics; Clobetasol; pimecrolimus

STUDY DESIGN:
Intervention Model Description: This study uses a three-arm, parallel assignment model comparing commonly used first-line therapies for vulvar lichen sclerosus. Participants are allocated into one of three non-randomized groups: (1) platelet-rich plasma (PRP) injections, (2) high-potency topical corticosteroid cream, or (3) topical calcineurin inhibitor. Each group receives a distinct intervention, and outcomes are assessed over 6 months using validated symptom and quality-of-life questionnaires and histopathological evaluation. The open-label design reflects real-world clinical practice and allows direct comparison of the effectiveness of each treatment modality.
Masking Description: This is an open-label study. No participants, care providers, investigators, or outcome assessors are masked to group assignment. No additional masking procedures are used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Platelet-Rich Plasma (PRP) Treatment (Experimental): Participants receive subcutaneous and submucosal injections of 5 ml autologous platelet-rich plasma (PRP) prepared using the Arthrex ACP Max™ system. PRP is injected into clinically affected vulvar areas and sites of itching or pain. Procedure performed once at study start. Outcomes are evaluated at baseline, 3 months, and 6 months; a vulvar biopsy is taken at 6 months.
  Interventions: Biological: Platelet-Rich Plasma (PRP) Treatment
- Topical High-Potency Corticosteroid (Active Comparator): Participants apply clobetasol propionate 0.05% cream (Dermovate) twice daily for the first 3 weeks and once daily for the following 3 weeks. Follow-up assessments occur at baseline, 3 months, and 6 months; a vulvar biopsy is taken at 6 months.
  Interventions: Drug: Clobetasol Propionate 0.05% Cream (Dermovate)
- Topical Calcineurin Inhibitor (Active Comparator): Participants apply pimecrolimus cream (Elidel) twice daily for 3 weeks and once daily for the following 3 weeks. Follow-up assessments occur at baseline, 3 months, and 6 months; a vulvar biopsy is taken at 6 months.
  Interventions: Drug: Pimecrolimus Cream (Elidel)

INTERVENTIONS:
Biological: Platelet-Rich Plasma (PRP) Treatment — Autologous platelet-rich plasma (5 ml) prepared using the Arthrex ACP Max™ Platelet-Rich Plasma System is injected subcutaneously and submucosally into clinically affected vulvar areas and sites of itching or pain. PRP is administered once at baseline following standard aseptic technique.
  Arms: Platelet-Rich Plasma (PRP) Treatment
Drug: Clobetasol Propionate 0.05% Cream (Dermovate) — Participants apply clobetasol propionate 0.05% cream topically twice daily for the first 3 weeks, followed by once daily for the next 3 weeks. This regimen represents standard high-potency corticosteroid therapy for vulvar lichen sclerosus.
  Arms: Topical High-Potency Corticosteroid
Drug: Pimecrolimus Cream (Elidel) — Participants apply pimecrolimus cream topically twice daily for 3 weeks, followed by once daily for the next 3 weeks. This regimen represents topical calcineurin inhibitor therapy for vulvar lichen sclerosus.
  Arms: Topical Calcineurin Inhibitor

SUMMARY:
Vulvar lichen sclerosus (VLS) is a chronic inflammatory skin condition that affects the vulvar area, often causing itching, burning, and pain, and may lead to scarring and narrowing of the vaginal opening. The condition significantly reduces the quality of life and may increase the risk of cancerous changes if left untreated.

This clinical study aims to evaluate and compare three commonly used treatment methods for women with biopsy-confirmed vulvar lichen sclerosus:

Topical corticosteroid therapy (clobetasol propionate 0.05%),

Topical calcineurin inhibitor therapy (pimecrolimus), and

Platelet-rich plasma (PRP) injections, which use the patient's own blood plasma rich in growth factors to support tissue healing.

A total of 45 participants aged 30 to 80 years will be enrolled and assigned to one of the three treatment groups. The effectiveness of therapy will be assessed using standardized questionnaires about symptoms and quality of life, as well as microscopic evaluation of tissue samples before and after treatment.

The study seeks to determine whether platelet-rich plasma (PRP) can serve as a safe and effective first-line treatment option for vulvar lichen sclerosus and to improve our understanding of the best therapeutic approaches for this chronic disease.

DETAILED DESCRIPTION:
Vulvar lichen sclerosus (VLS) is a chronic, progressive inflammatory dermatosis that primarily affects the skin and mucosa of the vulva and perineal region. The condition is most common in postmenopausal women and may cause severe itching, burning, pain during sexual intercourse, and, over time, scarring or anatomical changes that can significantly impair daily functioning and quality of life. If untreated, VLS may also increase the risk of developing vulvar intraepithelial neoplasia (VIN) or squamous cell carcinoma.

Despite the chronic nature of the disease, there is still no universally accepted standard of care for first-line treatment. Topical corticosteroids (such as clobetasol propionate 0.05%) are considered the mainstay of therapy, while topical calcineurin inhibitors (e.g., pimecrolimus or tacrolimus) are often used as alternatives or adjuncts in resistant cases. In recent years, regenerative methods such as platelet-rich plasma (PRP) therapy have emerged as a promising option. PRP is an autologous preparation containing a high concentration of platelets and growth factors that can stimulate tissue repair, reduce inflammation, and improve mucosal regeneration.

This open-label, non-randomized clinical study aims to evaluate and compare the therapeutic efficacy and safety of three treatment modalities in women with histopathologically confirmed vulvar lichen sclerosus:

PRP injection therapy using the Arthrex ACP Max™ Platelet-Rich Plasma System,

Topical corticosteroid therapy with clobetasol propionate 0.05% cream, and

Topical calcineurin inhibitor therapy with pimecrolimus cream.

A total of 45 participants will be recruited and assigned to one of the three treatment arms (15 per group). Clinical symptoms and quality of life will be evaluated using two validated questionnaires - the Vulvar Disease Symptom Score (VDSS) and the Dermatology Life Quality Index (DLQI) - at baseline, 3 months, and 6 months after treatment initiation. At the 6-month follow-up, a small biopsy from the vulvar area will be performed to assess histopathological changes, particularly the density of inflammatory cells.

The results of this study may help determine whether platelet-rich plasma (PRP) therapy could represent an effective and safe alternative to conventional topical treatments. Ultimately, this research could contribute to the development of more individualized and evidence-based therapeutic strategies for women suffering from vulvar lichen sclerosus.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 to 80 years.
2. Clinical diagnosis of vulvar lichen sclerosus confirmed by histopathological examination.
3. Ability and willingness to provide written informed consent for participation in the study.
4. Ability to comply with study procedures, including questionnaire completion and follow-up visits at baseline, 3 months, and 6 months.

Exclusion Criteria:

1. Lack of written informed consent to participate in the study.
2. Prior treatment for vulvar lichen sclerosus (any systemic or topical therapy targeted at VLS).
3. Current or past vulvar neoplasia, including vulvar intraepithelial neoplasia (VIN) or vulvar carcinoma.
4. Other organic or dermatologic causes of vulvar symptoms that could interfere with diagnosis or outcome evaluation.
5. Any condition that, in the opinion of the investigator, would interfere with study participation, follow-up, or accurate interpretation of results.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as women are eligible to participate, as the condition under study (vulvar lichen sclerosus) occurs exclusively in patients with vulvar anatomy.
Enrollment: 45 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in DLQI (Dermatology Life Quality Index) Score | Baseline, 3 months, 6 months
  The DLQI questionnaire assesses the impact of vulvar lichen sclerosus on patient quality of life. Scores range from 0 to 30, with higher scores indicating greater impairment. The study will measure the change in DLQI from baseline to 6 months across the three treatment groups.

SECONDARY OUTCOMES:
Change in VDSS (Vulvar Disease Symptom Score) | Baseline, 3 months, 6 months
  The VDSS evaluates symptom severity (itching, burning, pain, dyspareunia) associated with vulvar lichen sclerosus. The study assesses changes in total VDSS score over time to compare treatment effectiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinika Ginekologii i Ginekologii Onkologicznej, Szpital Uniwersytecki w Krakowie, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of vulvar biopsy samples and privacy considerations.